CLINICAL TRIAL: NCT03472157
Title: Prospective Multicentric, Open Label, Randomized Clinical Trial of Superiority, With Two Arms, Comparing Bariatric Surgery to the Recommended Medical Treatment for NASH
Brief Title: A Randomized Controlled Study Evaluating Bariatric Surgery as a Treatment for Severe NASH With Advanced Liver Fibrosis in Non-severe Obese Patients
Acronym: NASHSURG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016_78; 2017-A01575-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-02-13; First posted 2018-03-21 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Surgery; Obesity; NASH - Nonalcoholic Steatohepatitis; Cirrhosis
Keywords: Gastric bypass; Sleeve gastrectomy; Lifestyle therapy; NASH; Advanced fibrosis; Cirrhosis
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric surgery (Experimental): Two different types of bariatric surgery can be proposed: laparoscopic Roux-en-Y Gastric Bypass or a Laparoscopic sleeve gastrectomy.
  Decision of the surgery type will be made according to surgical expertise, habits of investigation centers and the patient's desire. All patients receive nutritional support and therapeutic education adapted to recommendations bariatric surgery care.
  Interventions: Procedure: Bariatric surgery
- Lifestyle therapy (Active Comparator): The group will received the medical standard treatment defined as lifestyle therapy combining diet with increased physical activity (standard treatment, control) (figure 1, design of study).
  Interventions: Other: Lifestyle therapy

INTERVENTIONS:
Other: Lifestyle therapy — Lifestyle habits (caloric intake and exercise) + pedometer
  Arms: Lifestyle therapy
Procedure: Bariatric surgery — Two different types of bariatric surgery can be proposed: laparoscopic Roux-en-Y Gastric Bypass or a Laparoscopic sleeve gastrectomy
  Arms: Bariatric surgery

SUMMARY:
The aim of the study is to demonstrate the superiority of bariatric surgery on the disappearance of NASH without worsening of fibrosis in comparison to medical standard treatment in obese patients (35 kg/m² > BMI ≥ 30 kg/m²) with NASH complicated of advanced fibrosis (F3 and F4 fibrosis grade according to Brunt score).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and agree to comply to the study protocol prior to enrolment.
* BMI and Brunt Fibriosis score:

  * For F3 fibrosis patients: 35>BMI≥ 30kg/m² ; Fibroscan ≥ 9kPa or FibrometreVM ≥0.526 predicting a F3 fibrosis score grade within 1 month before inclusion or F3 fibrosis score grade diagnosed by hepatic biopsy performed before inclusion.
  * For F4 fibrosis patients: 50>BMI≥ 30kg/m² ; Fibroscan ≥ 15kPa predicting a F4 fibrosis score grade within 1 month before inclusion or F4 fibrosis score grade diagnosed by hepatic biopsy performed before inclusion.
* Fibroscan ≥ 9kPa or FibrometreVM ≥0.526 predicting a F3 or F4 fibrosis score grade within 1 month before inclusion Or F3 or F4 fibrosis score grade diagnosed by hepatic biopsy performed before inclusion.
* Patient should agree to have one liver biopsy during the screening period (before randomization, the randomization will be permitted after at least a second reading performed by pathologist of CHRU Lille to confirm the histological diagnosis of NASH with advanced fibrosis (F3-F4)) for the diagnosis purpose (if no histological biopsy within 1 month before inclusion is available) and one at the end of the treatment period for assessment of the treatment effects.
* For patients with cirrhosis, patients must fulfil all the following criteria: Platelets > 125 000, PT > 80 %, Albumin > 35 g/L, MELD score at inclusion < 9, CPT score < 6, No history of previous decompensation, No oesophageal varices (endoscopy), No vascular shunt, ASA score ≤ III, Alcohol consumption lower than 20g/day for women and 30g/day for men.
* For hypertensive patients, hypertension must be controlled by stable dose of anti-hypertensive medication for at least 2 months prior to screening (and the stable dose can be maintained throughout the study).
* Female participating in the study must be either of non-child bearing (surgically sterilized at 6 month prior to screening or postmenopausal) or using an efficient contraception: hormonal contraception (including patch, contraceptive ring etc) intra-uterine device or other mechanical contraception
* Patient agrees to come to the study visits within the protocol-specified delay

Exclusion Criteria:

* Previous history of bariatric surgery (except gastric ring removed for more than 3 years).
* Decompensated cirrhosis (MELD> 7 CPT score> 5, previous history of decompensation (encephalopathy, ascites, jaundice, varicose vein rupture)
* Hepatocellular carcinoma
* Platelets <125 000; TP <80%; bilirubin <20 mmol / l; albumin <35 g / L.
* Other liver disease: alcohol consumption exceeding 20 g / day for women and 30g / day in men, HBV, HCV, CBP, CSP, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin.
* Being processed Cancer (chemotherapy, radiotherapy or hormone therapy)
* HIV positive patients
* Patients who had an acute cardiovascular episode, coronary Heart Disease (Angina pectoris, myocardial infarction, revascularization procedure), stroke or TIA (Transient Ischemic Attack) within the 6 months prior to screening Recent cardiovascular events (stroke, myocardial infarcts, etc…) in the past 6 months.
* Severe chronic respiratory disease.
* Severe chronic cardiac insufficiency (grade III and IV of NYHA classification).
* Pregnant or breastfeeding women.
* Simultaneous enrollment in another clinical trial.
* Drug abuse within the past year.
* Patient with contra-indication for bariatric surgery
* Gastic Banding, Biliopancreatic diversion and all the new bariatric surgery techniques are forbidden because the study design allow only the laparoscopic sleeve gastrectomy or laparoscopic Roux-en-Y gastric Bypaass.
* History of cancer, except:

  * Patients considered in remission for at least 5 years after onset of treatment.
  * Patients Treated and believed to be cured basal or squamous cell carcinoma of the skin or resected carcinoma of the cervix

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of disappearance of NASH without worsening of fibrosis grade | at 60 weeks after randomization
  Diagnosis of NASH on the liver biopsy

SECONDARY OUTCOMES:
Change in the NAS (Nafld Activity Score) score | at 60 weeks after randomization
  NAS is a histological score established on the liver biopsy. The NAS ranges form 0 to 8. 8 is associated with the highest severity.
Percentage of patients achieving at least a 2 point improvement in the NAS (≥2 points) without worsening of fibrosis grade | at 60 weeks after randomization
  NAS established on the liver biopsy
Change in the Brunt fibrosis score, | at 60 weeks after randomization
  Brunt fibrosis is a histological score ranges from 0 to 4. The Brunt fibrosis score is established on the liver biopsy. It is the recommended score for the evaluation of fibrosis in NASH and NAFLD. On the scale, "0" is an absence of fibrosis, whereas "4" matches with cirrhosis.
Change in the Metavir score | at 60 weeks after randomization
  METAVIR fibrosis score is established on the liver biopsy. METAVIR fibrosis is a histological score ranges from 0 to 4. This score is more discriminant than the Brunt score for the severe form of fibrosis that are included in this study.On the scale, "0" is an absence of fibrosis, whereas "4" matches with cirrhosis.
Change in the fibrosis area | at 60 weeks after randomization
  computerized morphometry analysis of fibrosis area
Change in the SF-36 quality of life score. | at 60 weeks after randomization
  SF-36 quality of life score
Percentage of patients with at least one of the following complications | through study completion
  complications: infection, thromboembolic complications, haemorrhage, rhabdomyolysis, hepatic decompensation and death
Percentage of patient achieving 5 and 10% of weight loss from randomization to end of treatment. | at 60 weeks after randomization
  Weight
Change in aspartate transaminase (AST) | at 60 weeks after randomization
  AST is a liver enzyme, used for the biological liver test evaluation.
Change in Alanine transaminase (ALT) | at 60 weeks after randomization
  ALT is a liver enzyme, used for the biological liver test evaluation.
Change in total bilirubin | at 60 weeks after randomization
  Total bilirubin is a liver enzyme, used for the biological liver test evaluation.
Change in GGT | at 60 weeks after randomization
  GGT (gamma glutamyl transferase) is a liver enzyme, used for the biological liver test evaluation. .
Change in ALP | at 60 weeks after randomization
  Alkalin Phosphatase is a liver enzyme, used for the biological liver test evaluation.
Change in INR (International Normalized Ratio) | at 60 weeks after randomization
  INR represents coagulation but also liver hepatocellular function.
Change in Albumin | at 60 weeks after randomization
  Albumin is used a marker of nutrition and hepatocellular function
Change in metabolic profile assessed by HOMA score | at 60 weeks after randomization
  HOMA is a score (scale) evaluating insulin resistance.
Change in Fasting glucose | at 60 weeks after randomization
  fasting glucose is a marker of diabetes and insulin resistance
Change in Glycated haemoglobin | at 60 weeks after randomization
  glycated haemoglobin is a surrogate marker for diabetes management and outcome.
Change in HDL cholesterol | at 60 weeks after randomization
  HDL cholesterol is a biomarker for lipid metabolism and cardiovascular risk
Change in serum triglycerides | at 60 weeks after randomization
  serum triglycerides is a biomarker for lipid metabolism and cardiovascular risk
Change in LDL cholesterol | at 60 weeks after randomization
  LDL cholesterol is a biomarker for lipid metabolism and cardiovascular risk
Change in total cholesterol. | at 60 weeks after randomization
  total cholesterol is a biomarker for lipid metabolism and cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mathurin, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHRU, Lille, France